CLINICAL TRIAL: NCT05484700
Title: SARS-CoV-2 Neutralizing Antibodies and Immunity After Vaccination of Recovered Patients With COVID-19 and Correlation With Immunity and Long-COVID-19 Symptoms
Brief Title: Antibodies and Immunity After Vaccination of Recovered Patients With COVID-19 and Long COVID-19 Symptoms
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Other Study IDs: 1013/2564(IRB3)
Record Dates: First submitted 2022-08-01; First posted 2022-08-02 (Actual); Last update posted 2022-08-05 (Actual); Status verified 2022-08

CONDITIONS: Long COVID-19
Keywords: Long COVID-19; antibody responsibility; immunogenicity
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Plasma Serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
We investigated the association between immune system responsibilities in Long COVID patients and Full recovery patients.

DETAILED DESCRIPTION:
This retrospective cohort study compared immunogenicity post COVID-19 between individuals (aged 18-65 years and had confirmed SARS-CoV-2 infection from January to May 2022 ) with residual Long COVID-19 symptoms (LC) and ones with full recovery (Full) related to pathophysiology, immunology and clinical consequence.

ELIGIBILITY:
Inclusion Criteria:

* Long COVID group; at longer than 1-month post COVID-19 based the presence of one of the three following symptoms: fatigue/myalgia, breathlessness, and anorexia
* Full recovery group; patients with asymptomatic symptoms
* post COVID-19 they had not received any additional COVID vaccine

Exclusion Criteria:

* people who received additional vaccination after leaving quarantine before the day of the immunization test
* pregnant patients,
* people who had a history of allergic reactions after COVID-19 vaccination or any drugs

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The COVID-19 patients who confirmed SARS-CoV-2 infection from January to May 2022 (during the Omicron wave), and post COVID-19 they had not received any additional COVID vaccine.
Sampling Method: Probability Sample
Enrollment: 305 (Estimated)
Dates: Start 2021-12-30 (Actual); Primary Completion 2022-07-25 (Actual); Study Completion 2022-12-29 (Estimated)

PRIMARY OUTCOMES:
Anti-SARS-CoV-2 RBD IgG | Baseline
  anti-SARS-CoV-2 receptor-binding domain immunoglobulin G(BAU/mL)
Anti-SARS-CoV-2 NP | Baseline
  surrogate Virus Neutralization Test (sVNT) (PRNT50 titer)
Microneutralization assays | Baseline
  Microneutralization assays using the authentic SARS-CoV-2 viruses

SECONDARY OUTCOMES:
Number of vaccine injection | Baseline
  Number of vaccine injection
Prevalence of Long COVID-19 symptoms | Baseline
  Number of participants with major Long COVID-19 symptoms including fatigue/myalgia, breathlessness, and anorexia by using the questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Korapat Mayurasakorn, MD., Principal Investigator — Doctor in Family Medicine
Locations (1):
- Faculty of Medicine Siriraj Hospital, Mahidol University, Bangkok Noi, Bangkok, Thailand